CLINICAL TRIAL: NCT02048644
Title: A Randomized, Double-blind, Placebo-controlled, Crossover Study to Assess the Effect of 28 Day Treatment With Fostair® Pressurized Metered-dose Inhaler (pMDI) 200/12 on Biomarkers of Platelet Adhesion in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Effect of Fostair® on Biomarkers of Platelet Adhesion in Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Acadmed18013
Record Dates: First submitted 2014-01-23; First posted 2014-01-29 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Platelets adhesion
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Beclomethasone; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo inhaler (Placebo Comparator): matched placebo inhaler, to be taken 2 puffs, twice a day for 28 days
  Interventions: Drug: placebo
- fostair (Experimental): fostair 100mcg/6mcg 2pufss, twice a day.
  Interventions: Drug: fostair

INTERVENTIONS:
Drug: fostair — beclometasone dipropionate 200mcg and formoterol 12 mcg delivered by inhaler, twice a day for 28 days
  Other Names: beclometasone dipropionate and formoterol fumarate
  Arms: fostair
Drug: placebo — placebo matched inhaler 2puffs to be taken twice a day for 28 days
  Arms: placebo inhaler

SUMMARY:
The investigator has recently studied markers of platelet activation in idiopathic pulmonary fibrosis (IPF) and found that in IPF patients there is a significantly increased platelet reactivity when compared with controls which is demonstrated by a concentration dependent increase in platelet-monocyte complex formation, platelet P-selectin expression and platelet fibrinogen binding in the presence of' the platelet agonists Adenosine diphosphate and L- Threonyl- L- phenylalanyl- L- leucyl- L- leucyl- L-argininamide (TFLLR).

During platelet activation the platelets degranulate releasing numerous profibrotic cytokines including Transforming growth factor beta and Platelet derived growth factor that are recognised to be important in the pathogenesis of IPF. It is therefore plausible that the observed increased platelet reactivity in IPF contributes to the fibrotic process through local activation and degranulation with release of proinflammatory and profibrotic mediators within the pulmonary circulation.

There is evidence that corticosteroid treatment may alter platelet adhesion, in a study of spontaneously hypertensive rat (SHR) increased circulating glucocorticoid, suppressed p-selectin expression. p selectin is a transmembrane protein present in the α granules of platelets. P selectin has a crucial role in platelet aggregation and platelet-leukocyte interactions, which are both potentially important mechanisms in the initiation and/or progression of tissue injury and development of thrombosis. In a study of patients with chronic obstructive pulmonary disease (COPD) exacerbation these were treated with either β agonists alone or β agonist and 40mg prednisolone and compared with a control group. At presentation the COPD patients had higher pulmonary artery pressure (PAP) higher p selectin and fibrinogen levels but lower Antithrombin III levels (AT III). The pulmonary artery pressure and fibrinogen levels were found to be significantly decreased in the steroid treated group whilst the p-selectin levels further increased in the non steroidal therapy patients.

Rationale for the Current Study

There is a significant unmet medical need for the treatment of IPF; the only medication approved for treatment of IPF in the United Kingdom (UK) is Pirfenidone and outside the UK there is none. The main goal of the current study is to evaluate the effect of Fostair on the biomarkers of platelet activation in IPF disease which the investigator believes play a pivotal role in the pathogenesis of IPF and whether this translates in to a clinically beneficial effect of Fostair on IPF disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects from 40 to 85 years of age
* Diagnosis of definite IPF according to American Thoracic Society / European respiratory symposium (ATS/ERS) Consensus Statement (2011) using either High-resolution computed tomography (HRCT) or surgical lung biopsy (SLB).
* Carbon monoxide transfer factor (TLco) of ≥ 30 % predicted ( historical measure accepted as long as within the last year).
* Able to maintain O2 saturation of ≥ 89% while breathing room air at rest.
* forced vital capacity (FVC) of 50-80% predicted value
* Negative serum pregnancy test at screening and negative urine pregnancy test at randomisation for female subjects of childbearing potential.
* Competency to understand the information given in the Ethics Committee approved Patient Information Sheet and Consent Form; subjects must sign the form prior to the initiation of any study procedures, unless the assessment is performed as standard of care for this disease

Exclusion Criteria:

* . Clinically significant respiratory diseases other than IPF, including asbestosis, other pneumoconiosis or hypersensitivity pneumonitis.

  * Clinically significant heart disease defined as a myocardial infarction documented by an ST elevation (STEMI) on electrocardiogram (ECG) within 6 months prior to screening, percutaneous coronary intervention or coronary artery bypass surgery within 6 months prior to screening, unstable angina pectoris, congestive heart failure (NYHA class III/IV or known left ventricular ejection fraction < 25%), ischaemic heart disease, right heart failure, significant right ventricular hypertrophy, or uncontrolled arrhythmia.
  * Current smokers
  * Use of any inhaled long acting beta-agonist or inhaled steroid within the 3 months prior to screening
  * Use of any medication to treat or possibly indicated in the treatment of IPF, such as pirfenidone, and oral corticosteroids.
  * Use of any Antiplatelet therapy which may alter assessment of study end points e.g. clopidogrel, Prasugrel, Dipyridamole etc.
  * History of cancer, precancerous state (eg, familial polyposis, breast cancer 1 (BRCA1),breast cancer 2 (BRCA2), carcinoma in-situ), other than non-melanomatous skin cancer, within 5 years prior to screening.
  * History or evidence of a clinically significant disorder, condition, or disease that, in the opinion of the investigator would pose a risk to subject safety or interfere with the study evaluations, procedures, or completion.
  * Participation in an investigational drug or device trial < 30 days prior to screening

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
platelet-monocyte complex formation | 1 month
  Measurements will include platelet-monocyte complex formation measured at baseline, and post investigational treatments at Visit 5 and visit 8.
platelet P-selectin expression | 1 month
  platelet p selectin expression will be measured at baseline, and post investigational treatments at Visit 5 and visit 8.
platelet fibrinogen binding | 1 month
  Platelet fibrinogen binding will be measured at baseline, and post investigational treatments at Visit 5 and visit 8.

SECONDARY OUTCOMES:
forced vital capacity | visit1, visit 5 and visit 8
  forced vital capacity will be measured at baseline and then at visit 5 and visit 8 following 1 months treatment of fostair or placebo
sputum eosinophils cells | 1 month
  inflammatory cells will be measured at baseline, and post investigational treatments at Visit 5 and visit 8.
six minute walk distance | 1 month
  six minute walk distance will be measured at baseline, and post investigational treatments at Visit 5 and visit 8.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Hart, MD, Principal Investigator — Hull University Teaching Hospitals NHS Trust
Locations (1):
- Respiratory Medicine Clinical trials Unit, Cottingham, East Yorkshire, United Kingdom

REFERENCES:
- [Result] Wright C, Arnell K, Fraser S, et al. S46 An RCT of 28 day treatment with Fostair® pMDI 200/12 BD on platelet biomarkers in patients with Idiopathic Pulmonary Fibrosis. Thorax 2015;70:A29-A30.
- See also: Publication Link — https://thorax.bmj.com/content/70/Suppl_3/A29.2